CLINICAL TRIAL: NCT00157625
Title: A Randomized Controlled Trial of Automatic Stop Orders for Urinary Catheterization in Hospitalized Patients
Brief Title: Automatic Stop Orders for Urinary Catheters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 03-24
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Urinary Tract Infections
Keywords: urinary infections, catheters, bacteriuria, trial
MeSH Terms: conditions — Urinary Tract Infections; Bacteriuria

INTERVENTIONS:
Behavioral: Automatic stop order

SUMMARY:
Urinary tract infections are the most common type of hospital-acquired infection. The majority of these infections result from the use of indwelling urinary catheters. Often caregivers leave them in unnecessarily. The purpose of this study is to assess the effectiveness of an automatic stop order (automatic removal or urinary catheters when they no longer needed) in reducing urinary infections.

DETAILED DESCRIPTION:
We will randomize patients with urinary catheters to either automatic stop orders or to usual care. The primary outcome will be urinary tract infection. Secondary outcomes will include days of indwelling urinary catheterization, symptomatic urinary tract infection, isolation of antimicrobial-resistant bacteria from catheterized urine, antimicrobial use, bacteremia (blood-stream) infection secondary to urinary tract infection, and cost. We hypothesize that use of the automatic stop order will significantly reduce hospital-acquired urinary tract infection.

ELIGIBILITY:
Inclusion Criteria:

* Urinary catheter for less than 48hrs

Exclusion Criteria:

* Patient with symptomatic urinary tract infection
* Latex allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630
Dates: Start 2003-04; Study Completion 2006-07

PRIMARY OUTCOMES:
Urinary tract infections

SECONDARY OUTCOMES:
days of indwelling urinary catheterization,
symptomatic urinary tract infection,
isolation of antimicrobial-resistant bacteria from catheterized urine,
antimicrobial use,
bacteremia (blood-stream) infection secondary to urinary tract infection,
cost

CONTACTS AND LOCATIONS:
Overall Officials: Mark B Loeb, MD MSc FRCPC, Principal Investigator — McMaster University
Locations (3):
- Canada (3):
  - McMaster University Medical Centre, Hamilton, Ontario
  - Henderson Hospital, Hamilton, Ontario
  - Hamilton General Hospital, Hamilton, Ontario

REFERENCES:
- [Derived] Ellahi A, Stewart F, Kidd EA, Griffiths R, Fernandez R, Omar MI. Strategies for the removal of short-term indwelling urethral catheters in adults. Cochrane Database Syst Rev. 2021 Jun 29;6(6):CD004011. doi: 10.1002/14651858.CD004011.pub4. PMID 34184246